CLINICAL TRIAL: NCT03668327
Title: Preterm Birth Cohort Study in Guangzhou
Acronym: PBCSG
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018090501
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Neurodevelopment; Immune Development; Host and Microbiome
Keywords: Preterm; Cohort; Early development; Child
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At delivery: maternal blood, cord, cord blood and placenta. During infancy: dry blood spot, stool and blood. During childhood: blood, buccal swab and stool.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The Preterm Birth Cohort Study in Guangzhou (PBCSG) aims to explore the impact of genetic and environmental factors including life styles on preterm birth, to examine the interaction effect between these factors, and to follow up the short-term and long-term outcomes of preterm childrens.

DETAILED DESCRIPTION:
Preterm birth has become the leading cause of neonatal death and the second leading cause of death among children under five years of age. Preterm childrens are more susceptible to adverse health problems including brain injury and neurodevelopment delay, and are at risk of chronic diseases which could impair the health status and life quality later in life. However, the causes of preterm birth is still not clear, and there are no effective prediction and preventive strategies. The Preterm Birth Cohort Study in Guangzhou (PBCSG) will collect the epidemiological,clinical information and biological specimens including maternal blood,cord blood, placenta, children's blood and stool samples of preterm childrens and their mothers. More importantly, childrens' health status, physical and neurodevelopment will be followed up to late childhood and adolescence. The preterm birth cohort would help to explore the mechanism of preterm birth and to examine the short- and long-term influence of preterm birth on physical health and neurodevelopment of childrens.

ELIGIBILITY:
Inclusion Criteria:

1. Born before 37 weeks of gestation
2. Born in Guangzhou Women and Children's Medical Center
3. Intended to remain in Guangzhou for more than 3 years

Exclusion Criteria:

1. Multiple birth
2. Stillbirth
3. With major congenital abnormalities

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population are childrens born before 37 weeks of gestation and their mothers in Guangzhou.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopment at early childhood | At age of 1 year
  Assessed by using the Gesell Developmental Schedules, which include adaptive, gross motor, fine motor, language, and social function domains. Higher score in each domain is considered a better outcome, while no more than 85 is defined as suspected development retardation

SECONDARY OUTCOMES:
Intelligence quotient of offspring | At age of 6 years old
  Assessed by using Wechsler's Intelligence Scale for Children (WISC), which can generate a full scale intelligence quotient score and five primary index scores including verbal comprehension, visual spatial, fluid reasoning, working memory, and processing speed. Intelligence quotient ranges from 40 to 160,in which less than 70 is defined as mental retardation
Height changes during childhood and adolescence | At birth, age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 year
  Measured by nurses in clinic using a standard tool
Weight changes during childhood and adolescence | At birth, age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 year
  Measured by nurses in clinic using a standard tool
Change of intestinal flora during early childhood | At age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
  Assessed by analyses of stool samples
Changes of body fat percentage during early childhood | At age of 3 years, 6 years, 12 years and 18 years old
  Assessed by Dual Energy X-Ray Absorptiometry (defined as total mass of fat divided by total body mass)
Changes of bone density during early childhood | At age of 3 years, 6 years, 12 years and 18 years old
  Assessed by Dual Energy X-Ray Absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, MD,PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, China, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694